CLINICAL TRIAL: NCT06818071
Title: Application of Gamified Elements to Increase Daily Step Count in University Students in Taiwan A Randomized Controlled Trial
Brief Title: Using Gamified Elements to Increase Daily Step Count in University Students in Taiwan A RCT
Acronym: AGEPATWRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Jeffrey Zen Liu, PhD Candidate, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N202310009; N2023100009 (Other: TAIPEI MEDICAL UNIVERSITY INSTITUTIONAL REVIEW BOARD)
Record Dates: First submitted 2025-01-17; First posted 2025-02-10 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Physical Activity; Gamification; Daily Step Count
Keywords: Gamified Elements; Gamification; Daily Step Count; Phsyical Activity; Health Promotion; Behavioral Change
MeSH Terms: conditions — Motor Activity | interventions — Intersectoral Collaboration

STUDY DESIGN:
Intervention Model Description: Participants are randomized into four different groups: 1. Control, 2. Individual Gamified Elements Group (IGG), 3. Combined Gamified Elements Group (CGG), and 4. Explicit Gamification Group (EGG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Participants in this group will not interact with the study during the study period, but will complete body measurements and questionnaires at Week 1, 9, and 12 and provide weekly daily step count averages for the study period.
- Individual Gamified Elements Group (IGG) (Experimental): IGG Participants interact with each gamified element one by one. They will will set a daily step goal after developing a baseline during the first week. During the subsequent weeks, IGG participants will receive health information on a daily basis (Week 2), gain points for a 7-11 gift card (Week 3), compete with their group on a leaderboard (Week 4), group up with other IGG participants and compete with other groups (Weeks 5 & 6), then play a mobile game that focuses on explicit gamification (Pikmin Bloom, Weeks 7 & 8). IGG Participants will complete the TANITA body measurement, blood pressure & heart rate, waist & hip circumference, and the questionnaire at Weeks 1, 9, & 12.
  Interventions: Behavioral: Points and Leaderboards; Behavioral: Social Aspects; Behavioral: Health Messages; Behavioral: Pikmin Bloom
- Combined Gamified Elements Group (CGG) (Experimental): CGG Participants interact with gamified element by adding additional ones each week. They will will set a daily step goal after developing a baseline during the first week. During the subsequent weeks, ICGG participants will receive health information on a daily basis (Week 2-8), gain points for a 7-11 gift card (Week 3-8), compete with their group on a leaderboard (Week 4-8), group up with other IGG participants and compete with other groups (Weeks 5-8), then play a mobile game that focuses on explicit gamification (Pikmin Bloom, Weeks 7-8). CGG Participants will complete the TANITA body measurement, blood pressure & heart rate, waist & hip circumference, and the questionnaire at Weeks 1, 9, & 12.
  Interventions: Behavioral: Points and Leaderboards; Behavioral: Social Aspects; Behavioral: Health Messages; Behavioral: Pikmin Bloom
- Explicit Gamified Elements Group (EGG) (Experimental): EGG Participants interact with each gamified element one by one. They will will set a daily step goal after developing a baseline during the first week. During the subsequent weeks, EGG participants will play a mobile game that focuses on explicit gamification (Pikmin Bloom, Weeks 2-8). EGG Participants will complete the TANITA body measurement, blood pressure & heart rate, waist & hip circumference, and the questionnaire at Weeks 1, 9, & 12.
  Interventions: Behavioral: Pikmin Bloom

INTERVENTIONS:
Behavioral: Points and Leaderboards — Participants will have the opportunity to gain points if they meet their self-set daily step goal throughout the experiment period.
  Participants will also compete with others in their own respective groups on a leaderboard in regards to each day's daily step count.
  Other Names: PBLs
  Arms: Combined Gamified Elements Group (CGG); Individual Gamified Elements Group (IGG)
Behavioral: Social Aspects — Participants will be randomly assigned into groups of three to compete with other groups based on their daily step count. Each day, one participant will be randomly selected to represent the group against their opponent. If they walked more than their randomly selected opponent, the participant's group will receive a positive, encouraging message congratulating them for winning that day. If they did not walk more than their randomly selected opponent, they will receive a motivational message to encourage them to walk more.
  Other Names: Collaboration; Competition; Teamwork
  Arms: Combined Gamified Elements Group (CGG); Individual Gamified Elements Group (IGG)
Behavioral: Health Messages — Experiment participants will receive messages that encourage healthy behaviors. These include topics such as: nutrition, sleep, physical activity, and decreased consumption/use of unhealthy products (tobacco, alcohol, etc.).
  Arms: Combined Gamified Elements Group (CGG); Individual Gamified Elements Group (IGG)
Behavioral: Pikmin Bloom — Participants will play the mobile game Pikmin Bloom, which encourages users to increase their daily step count and allows them to utilize various gamified elements to do so. The game has many gamified elements included, such as personalization and avatar, social aspects, competition, collaboration, progression, and many more.
  Other Names: Explicit Gamification; Mobile gaming
  Arms: Combined Gamified Elements Group (CGG); Explicit Gamified Elements Group (EGG); Individual Gamified Elements Group (IGG)

SUMMARY:
Background: Physical inactivity is a major factor in the onset of non-communicable diseases (NCDs) worldwide. Heart disease, Diabetes mellitus, and hypertensive diseases are among the top 10 leading causes of death in Taiwan in 2021. Although 81.6% of Taiwanese participants in a 2022 nationwide survey responded that they exercised regularly, the Health Promotion Administration stated that 50.3% of the population from 2017-2020 is overweight or obese, up from 32.7% in 1993-1996. The intention-behavior gap in habit formation is difficult to overcome for most, especially when self-motivation is the biggest factor. Gamification, the use of game elements in non-game settings, and game elements can be used to lower the bar necessary for individuals to develop healthier daily habits.

Aim: This study aims to investigate the effects of applying gamified elements on the daily lives of university students in Taiwan to increase their daily step count as compared to their baseline and the control group, along with changes in certain health indicators, overall physical activity, sleep behavior & quality, and mental health, whether combining gamified elements is more effective than implementing gamified elements individually, and if implicit or explicit gamification is more effective.

Methods: 255 participants were recruited and, after providing informed consent, randomized into four groups: (1) Control, (2) Individual Gamified Elements Group (IGG), (3) Combined Gamified Elements Group (CGG), and (4) Explicit Gamification Group (EGG). Control group participants will add the official LINE account, submit weekly summaries of their DSC and to complete the three questionnaires. IGG, CGG, and EGG participants will be asked to add the official LINE account, download Google Fit onto their smartphone, establish a baseline for the first seven days, then set a Daily Step Count Goal (DSG) of an increase of 25%, 33%, or 50% on Day 7 of the study. IGG and CGG participants will then engage in various interventions, including Nudging (Week Two), and gamified interventions, including Points, Badges, & Leaderboards (PBLs) (Weeks Three & Four), Social Aspects (Weeks Five and Six), and Personalized Avatar & Progression via Explicit Gamification (Weeks Seven & Eight). IGG participants will engage with the multiple forms of gamified elements separately throughout the experiment, while CGG participants will slowly combine gamified elements as the experiment progresses (i.e. Week 2 Nudging, Week 3 Nudging + Points, Week 4 Nudging + Points + Leaderboard, etc.). EGG Participants will play Pikmin Bloom, which includes various gamified elements, for the duration of the study (8 weeks). Participants will complete the questionnaire at three points: the beginning of the experiment (initial check-in), the end of the experiment (8 weeks), and at follow-up (twelve weeks). The primary aim will be to determine whether or not the implementation of gamified elements will lead to an increase in overall DSC from baseline to 8 and 12 weeks, along with a certain percentage of patient-days that self-set DSGs are met at 8 and 12 weeks, as compared to the control group. Secondary outcomes include: how increasing participants' DSC will affect their health indicators, physical activity, mental health, and sleep behavior & quality, comparing the effectiveness of combined gamified elements vs. individual gamified elements in increasing participants' DSC, and if implicit or explicit gamification is more effective at increasing DSC.

DETAILED DESCRIPTION:
The purpose of this study is to measure the effects of the application of gamified elements on the intervention participants' daily step count (DSC) as compared to their baseline and control group. Potential candidates for the study will provide informed consent after being informed of the study, answer the questionnaire (consisting of the International Physical Activity Questionnaire - Short Form (IPAQ-SF), Pittsburgh Sleep Quality Index -Chinese version (PSQI-C), Insomnia Severity Index - Chinese Version (ISI-C), and the 12-item Short Form Survey (SF-12)). Participants will also measure their Blood Pressure, Heart Rate, Body Mass Index (BMI), Waist-to-Hip Ratio (WHR), Body Fat Percentage, Muscle Mass, Bone Density, and Body Fluid Amount. Intervention participants will establish a baseline for the first seven days, then set a Daily Step Goal (DSG) of an increase of 25%, 33%, or 50%. IGG and CGG participants will then engage in various interventions, including Nudging (Week Two), and gamified interventions, including Points, Badges, & Leaderboards (PBLs) (Weeks Three & Four), Social Aspects (Weeks Five and Six), and Personalized Avatar & Progression (Weeks Seven & Eight). Points accumulated will be reset each week to give participants a fresh start. EGG participants will play Pikmin Bloom for the study duration. The primary aim will be to determine whether or not the implementation of gamified elements will lead to an increase in overall DSC from baseline to 8 and 12 weeks, along with a certain percentage of patient-days that self-set DSGs are met at 8 and 12 weeks, as compared to the control group. Secondary outcomes include: how increasing participants' DSC will affect their health indicators, physical activity, mental health, and sleep behavior & quality, comparing the effectiveness of combined gamified elements vs. individual gamified elements in increasing participants' DSC, and if implicit or explicit gamification is more effective at increasing DSC.

Two previous studies conducted in the United States of America are the main basis for this study. The first study, "Effectiveness of Behaviorally Designed Gamification Interventions with Social Incentives for increasing Physical Activity Among Overweight and Obese Adults Across the United States - The STEP UP Randomized Clinical Trial", published in 2019 by Mitesh S. Patel et al, found that using gamified interventions - support, collaboration, and competition - "significantly increased physical activity compared with the control group during the 24-week intervention".

The second study, "Effect of Behaviorally Designed Gamification with Social Incentives on Lifestyle Modification Among Adults with Uncontrolled Diabetes - A Randomized Clinical Trial", published in 2021 by Mitesh S. Patel et al, found that gamified interventions "designed to enhance support or competition each significantly increased physical activity relative to controls during the 1-year intervention".

Potential risks in this study will be minimal and the risk/benefit ratio will be in favor of the participants. To reduce the potential of unexpected adverse events, the research team will assess the potential participants at the initial check-in to the best of their ability on their potential to complete the experiment. If participants are deemed unfit to complete the experiment (injury, unable to participate for 12 weeks, etc.), the research team will inform the participant and remove them from the study.

This study is based on studies conducted in the United States mentioned in Section 2.3 that have resulted in some significant results in certain vulnerable populations. The research team wanted to conduct a study in the similar vein but with alterations in regards to the overall concepts and population. The study population investigated in this study will be different but the hope of this research is that if there is significance in the application of gamified elements on the increase of DSC, then we will be able to conduct further studies in different populations, including vulnerable ones, to improve health and healthy behaviors.

This study will be conducted in compliance with the protocol approved by the Institutional Review Board, and according to Good Clinical Practice standards. No deviation from the protocol will be implemented without the prior review and approval of the IRB except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the IRB as soon as possible.

255 participants from Taipei Medical University ages 18 to 35 enrolled, have access to a smartphone, and have a LINE account were enrolled in the study. The researchers will use convenience sampling to enroll participants into the study.

The purpose of this study is the explore the potential effectiveness of the application of gamified elements to promote physical activity among university students in Taiwan.

Research objectives of this study are to:

1. Determine whether or not the implementation of gamified elements will lead to an increase in overall DSC from baseline to 8 and 12 weeks, along with a certain percentage of patient-days that self-set DSGs are met at 8 and 12 weeks, as compared to the control group.
2. Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators, mental health, and sleep behavior and quality
3. comparing the effectiveness of combined gamified elements vs. individual gamified elements in increasing participants' DSC, and
4. Determine the potential effectiveness of utilizing implicit gamification compared to explicit gamification and their effects on increasing DSC and percentage of meeting DSGs.

This will be a randomized controlled trial. The study recruited 255 participants from Taipei Medical University and randomly distribute them into four groups by having them pick a unique number from a bowl: (1) control, (2) individual gamified elements group, (IGG), (3) combined gamified elements group (CGG), and (4) Explicit Gamification Group (EGG). Informed consent will be collected. The study will take measurements at three points in time: (1) the initial check-in, (2) end of the experiment (8 weeks), and (3) one-month follow-up (12 weeks). These measurements include blood pressure, heart rate, Body Mass Index (BMI), Waist-to-Hip Ratio (WHR), Body Fat Percentage, Muscle Mass, Bone Density, Body Fluid Amount, and answering a questionnaire consisting of International Physical Activity Questionnaire - Short Form (IPAQ-SF), Pittsburgh Sleep Quality Index - Chinese version (PSQI-C), Insomnia Severity Index - Chinese Version (ISI-C), and the 12-item Short Form Survey (SF-12).

The experimental period of the study will last 8 weeks with a 4-week follow-up, for a total of 12 weeks. After completing the initial check-in and submitting their informed consent forms, participants will be asked to download Google Fit (if they don't already have the app installed) and add the study's official LINE account.

Control group participants will be prompted at the end of the experiment (Week 8) to submit a screenshots of their weekly averages of their DSC from Google Fit. This, along with the questionnaire portions (at Weeks 8 and 12), will be the only time that the research team will contact the control group.

For the first week of the study, the IGG, CGG, and EGG participants will be asked to develop a baseline of their daily step count (DSC). Participants will not be contacted or reminded to meet any certain DSC during this period of seven days. After the first week, the research team will contact the participants and ask them to submit their weekly DSC average (found in Google Fit) and establish a self-set daily step count goal (DSG), which will be an increase of 25%, 33%, or 50% of baseline - for at least an increase of 1,000 steps.

For the second week of the study, the research team will utilize nudging to remind participants to meet their self-set DSGs. The official LINE account will send two messages per day at 10 AM and 7 PM as a reminder to meet their DSGs - the morning message will be a more generalized message while the nighttime message will include a reminder to submit a screenshot of their daily step count via Google Fit - the study's way of monitoring the participants' DSC and DSGs.

For the rest of the experiment, EGG participants will download Pikmin Bloom and Pokémon Sleep, and play the games for the duration of the study period. The games will be explained below.

For the third week of the study, the research team will notify the IGG and CGG participants to meet their DSGs to gain points towards an additional financial incentive at the end of the study. Participants can gain a total of 70 points each week (10 points per day) if they meet their DSGs, and will not gain points if they fail to meet their DSGs. Starting from this section, the IGG and CGG will begin to differentiate, with the IGG not receiving the nudging messages from the previous week and the CGG continuing to receive messages until the end of the study. CGG participants will also be eligible for further weekly financial incentives if they meet their weekly goals for the rest of the study for up to a total of $1,000 NTD; their points will be reset at the beginning of each week.

For the fourth week of the study, a leaderboard will be used. IGG and CGG participants will begin competing against each other within their designated groups (e.g. IGG participants will compete with each other, CGG participants will compete with each other). A leaderboard will be updated daily at noon and include participants' daily step count over the week. Participants will be reminded to submit their DSC or risk losing points for that day. CGG participants will continue to receive daily notifications twice a day; points will also be reset this week to emulate the fresh start theory.

For the fifth and sixth week of the study, IGG and CGG participants will be placed into groups of three and randomly selected to compete with another team within their intervention clusters. We will use an online software (https://www.randomlists.com/team-generator) to randomize the 60 participants into 20 groups. They will face different teams during the two weeks. This section will emulate social aspects, as participants will have to collaborate within their team while also competing against other participants. One participant within each group will be randomly selected each day to represent the group; therefore, this promotes communication and collaboration among group members to encourage each other to meet their DSGs to gain points. Teams will be notified at the beginning of each day whether or not their opponents have met their DSGs and gained points. The CGG participants will continue receiving notifications daily, along with gaining points for their individual goal and also competing against everyone on the leaderboard.

For the seventh and eighth week of the study, participants will be asked to download a mobile game - Pikmin Bloom - to assist in meeting their DSGs.

Pikmin Bloom is a mobile application focused on increasing the user's daily step count via personalized avatar, progression, and various in-game rewards. The game will tie into the user's smartphone's native health application (Apple Health for iOS or Google Fit for Android) and link the daily step count to the game. The game provides a daily summary of the user's steps at night, which helps users reflect on their DSC.

Participants will create an account and be asked to interact with the games. Pikmin Bloom will track their daily steps. Participants will use Pikmin Bloom to track their steps and submit their DSC screenshot to the research team from within the mobile game instead of a screenshot of Google Fit. Participants can create an avatar and will progress towards certain goals given within the game. The game is mainly based on DSC and players progress when certain goals are achieved via DSC. IGG participants will be tasked with submitting a screenshot of the in-game DSC screen. CGG participants will also submit screenshots of their DSC via Pikmin Bloom, alongside receiving notifications, points, monitoring the daily leaderboard, and competing against their randomly assigned opponents.

After the conclusion of the experiment, participants will be asked to come in to complete the second questionnaire and measurements. The research team will remind them that a follow-up will be performed four weeks from the end of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Taipei Medical University student
* Ages 18 - 35
* Access to smartphone
* LINE messaging account
* Provide Informed Consent

Exclusion Criteria:

* Not currently participating in other studies regarding health
* Cannot commit to the entire study period (12 weeks)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Increase Daily Step Count and Daily Step Goals Met with Gamified Elements | 12 weeks (8 week experiment, 4 week follow-up)
  Determine whether or not the implementation of gamified elements will lead to an increase in overall DSC from baseline to 8 and 12 weeks, along with a certain percentage of patient-days that self-set DSGs are met at 8 and 12 weeks, as compared to the control group.

SECONDARY OUTCOMES:
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. Blood Pressure (systolic and diastolic blood pressure in mmHg) will be measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. The study will evaluate the participants' Heart Rate (beats per minute) at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. Body mass index (BMI, weight and height will be combined to report BMI in kg/m^2) will be measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. Waist-to-Hip Ratio (WHR, waist circumference and hip circumference will be combined - [Waist Circumference/Hip Circumference] - to report WHR) measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. Body Fat Percentage will be evaluated using a TANITA body measurement machine and measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. Muscle Mass (kg) will be evaluated using a TANITA body measurement machine and measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. Total Body Water Percentage will be evaluated using a TANITA body measurement machine and measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on health indicators. Bone Density (kg) will be evaluated using a TANITA body measurement machine and measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up).
Potential Effectiveness of Increased DSC on health indicators | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on overall physical activity. The International Physical Activity Questionnaire-Short Form (IPAQ-SF) will be administered at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up). The seven-item self-reported questionnaire asks about physical activity (vigorous, moderate, and walking) and amount of sitting in the past seven days.
Effectiveness of Individual Gamified Elements vs. Combined Gamified Elements | 12 weeks (8 week experiment, 4 week follow-up)
  IGG participants will interact with gamified elements on an individual basis, while CGG participants will gradually accumulate more gamified elements as the experiment continues. The research team would like to evaluate the effects of these gamified elements on the participants' DSC throughout the experiment period and evaluate whether or not the accumulation of gamified elements increases participant DSC as compared to gamified elements being implemented one at a time.
Implicit vs. Explicit Gamification Effect on Participant DSC | 12 weeks (8 week experiment, 4 week follow-up)
  Evaluate the effectiveness of implicit gamification (research team-designed gamified elements like points, leaderboards, and social aspects) vs. explicit gamification (Pikmin Bloom mobile game) and their effects on participant DSC over the experiment period.
Potential Effectiveness of Increased DSC on sleep behavior and quality | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on sleep behavior and quality. Sleep behavior and quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI) questionnaire and measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up). The 19-question self-reported questionnaire evaluates sleep quality and sleep disturbances in the past 30 days.
Potential Effectiveness of Increased DSC on sleep behavior and quality | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on sleep behavior and quality. Sleep behavior and quality will be evaluated using the Insomnia Severity Index (ISI) questionnaire and measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up). The 7-question self-report questionnaire evaluates aspects of insomnia, including: difficulty falling asleep, difficulty staying asleep, problems with waking up too early, satisfaction with current sleep pattern, interference of sleep problems with daily functioning, noticeability of sleep problems by others, and distress caused by sleep problems.
Potential Effectiveness of Increased DSC on mental health and well-being | 12 weeks (8 week experiment, 4 week follow-up)
  Determine the potential effectiveness of increasing participants' DSC and its effects on mental health. Mental health and well-being will be evaluated with the 12-item Short Form Survey (SF-12), and measured at 3 different times: 1) Week 1 (Start of Experiment), Week 9 (Experiment End), and Week 12 (Follow-Up). The 12-item self-report survey designed to evaluate an individual's physical and mental health. It provides two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Jen Tsai, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yao J, Lim N, Tan J, Matthias Muller A, Martinus van Dam R, Chen C, Tan CS, Muller-Riemenschneider F. Evaluation of a Population-Wide Mobile Health Physical Activity Program in 696 907 Adults in Singapore. J Am Heart Assoc. 2022 Jun 21;11(12):e022508. doi: 10.1161/JAHA.121.022508. Epub 2022 Jun 14. PMID 35699174
- [Background] Agarwal AK, Waddell KJ, Small DS, Evans C, Harrington TO, Djaraher R, Oon AL, Patel MS. Effect of Gamification With and Without Financial Incentives to Increase Physical Activity Among Veterans Classified as Having Obesity or Overweight: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2116256. doi: 10.1001/jamanetworkopen.2021.16256. PMID 34241628
- [Background] Fanaroff AC, Patel MS, Chokshi N, Coratti S, Farraday D, Norton L, Rareshide C, Zhu J, Szymczak JE, Russell LB, Small DS, Volpp KGM. A randomized controlled trial of gamification, financial incentives, or both to increase physical activity among patients with elevated risk for cardiovascular disease: rationale and design of the be active study. Am Heart J. 2023 Jun;260:82-89. doi: 10.1016/j.ahj.2023.02.014. Epub 2023 Mar 2. PMID 36870551
- [Background] Patel MS, Small DS, Harrison JD, Hilbert V, Fortunato MP, Oon AL, Rareshide CAL, Volpp KG. Effect of Behaviorally Designed Gamification With Social Incentives on Lifestyle Modification Among Adults With Uncontrolled Diabetes: A Randomized Clinical Trial. JAMA Netw Open. 2021 May 3;4(5):e2110255. doi: 10.1001/jamanetworkopen.2021.10255. PMID 34028550
- [Background] Patel MS, Small DS, Harrison JD, Fortunato MP, Oon AL, Rareshide CAL, Reh G, Szwartz G, Guszcza J, Steier D, Kalra P, Hilbert V. Effectiveness of Behaviorally Designed Gamification Interventions With Social Incentives for Increasing Physical Activity Among Overweight and Obese Adults Across the United States: The STEP UP Randomized Clinical Trial. JAMA Intern Med. 2019 Dec 1;179(12):1624-1632. doi: 10.1001/jamainternmed.2019.3505. PMID 31498375
- [Derived] Liu JZ, Yu Chen R, Rouyard T, Munkhtogoo D, Tsai FJ. Effects of Different Gamification Delivery Strategies on Physical Activity in Young Adults: A Randomized Controlled Trial. Am J Prev Med. 2026 Feb 6:108297. doi: 10.1016/j.amepre.2026.108297. Online ahead of print. PMID 41655647